CLINICAL TRIAL: NCT01516125
Title: Screening of Healthy Adults for Genetic Variations That Control Fatty Acid Processing
Status: Completed | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH); Office of Dietary Supplements (ODS) (NIH); University of Arizona (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00016822; P50AT002782 (NIH)
Record Dates: First submitted 2012-01-11; First posted 2012-01-24 (Estimated); Last update posted 2023-11-30 (Actual); Status verified 2023-03

CONDITIONS: Healthy
Keywords: healthy adult; genetic variation; botanical oils; polyunsaturated fatty acid; fish oil; fat metabolism; Genetic variation of fat metabolism in healthy adults

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — A small saliva sample for screening purposes will be collected. If documentation from a personal physician of blood glucose and lipid levels are unavailable, we will collect a small tube (10-12 ml) of blood to determine these measurements.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Screening only - no intervention

SUMMARY:
The purpose of this research study is to screen healthy African American and Caucasian persons for specific differences in genes that control how fats are processed in the body.

DETAILED DESCRIPTION:
Healthy African American and Caucasian persons will be screened for specific differences in genes that control how fats are processed in the body. Persons with the needed genotypes will be added to a database of healthy persons who may be asked to join a larger study comparing differences in diet on lipid metabolism and inflammatory biomarkers as well as future studies. A key hypothesis for the larger study is that variations in genes involved in lipid metabolism play a role in determining levels of long chain polyunsaturated fatty acids (LC-PUFAs).

ELIGIBILITY:
Inclusion Criteria:

* Be Caucasian or African American between 21-65 years of age
* Be healthy and free of any major illness
* Be a nonsmoker
* Have an intact gallbladder
* Have TG < 150 and blood pressure less than 130/90
* Must be willing to be re-contacted for future studies

Exclusion Criteria:

* Not have: myocardial infarction, vascular surgery or stroke within the past year
* Not be taking niacin, more than 100 mg aspirin/day or montelukast allergy medications
* BMI equal to or greater than 30 or less than 19
* Fasting glucose greater than 125 mg/dl
* Pregnancy

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Caucasian or African American adults between 21 and 65 years of age
Sampling Method: Non-Probability Sample
Enrollment: 458 (Actual)
Dates: Start 2011-09 (Actual); Primary Completion 2019-04-17 (Actual); Study Completion 2019-04-17 (Actual)

PRIMARY OUTCOMES:
Determine the genotype at the rs174537 single-nucleotide polymorphism (SNP) in the fatty acid desaturate (FADS) gene cluster | up to 52 months

CONTACTS AND LOCATIONS:
Overall Officials: Susan Sergeant, Ph.D., Principal Investigator — Wake Forest University Heath Sciences
Locations (1):
- Wake Forest Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
This is a screening (one visit) to recruit healthy people for genotyping and re-contact for future studies